CLINICAL TRIAL: NCT03846674
Title: Depression Symptoms Among Ever Married Females Attending Primary Health Care Units in Dairut City
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MFMukhtar, principal investigator, Assiut University
Other Study IDs: 17100426
Record Dates: First submitted 2019-02-10; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depression is defined as a cluster of specific symptoms with associated impairment. The clinical and diagnostic features of the disorder are broadly similar in adolescents and adults.

Nevertheless, depression in adolescents is more often missed than it is in adults, possibly because of the prominence of irritability, mood reactivity, and fluctuating symptoms in adolescents.

While depression is the leading cause of disability for both males and females, the burden of depression is 50% higher for females than males. In fact, depression is the leading cause of disease burden for women in both high-income and low- and middle-income countries.

DETAILED DESCRIPTION:
The prevalence of depression in children is low (<1% in most studies) with no sex differences, and then rises substantially throughout adolescence.

Okasha found that the lifetime prevalence of depression in urban and rural Egyptian populations to be 11.4 and 19.7% Several studies show that depression during adolescence is a risk factor of academic failures, marriage struggles, suicide attempts, interpersonal conflicts, unemployment, drug abuse; it is also a strong predictor of adulthood depression.

Girls married too early are also more likely to experience domestic violence, abuse and forced sexual relations.

Similarly early married females when interact with new individuals after marriage are unable to deal them psychologically which is mostly due to the bad behaviours shown from in-laws towards them thus leading to lower self-esteem, increasing their risk of clinical depression which on extreme aspect can cause suicidal attempts.

ELIGIBILITY:
Inclusion Criteria:

* Married
* Divorced
* Separated
* Widow

Exclusion Criteria:

* Cases diagnosed with mental disorders
* History of mental disorders
* Family history of mental disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The city has a total population of 92144 and total numbers of families 20942.There are two primary health care centers in Dairut city that provide the primary care services.
  * Medical Centre (MC) covers the Eastern part of Dairut City.
  * Maternal and child care center west Dirout (MCCC) covers the Western part of the city.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-12-22 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms among ever married females attending primary health care units in Dairut City | 6 months
  All recruited women will complete a structured self-administered questionnaire which will include:
  Socio-demographic variables: , age for wife, age for husband, residence, education for wife, education for husband, occupation for wife, occupation for husband, parity.
  The Patient Health Questionnaire (PHQ) is a new instrument for making criteria-based diagnoses of depressive and other mental disorders commonly encountered in primary care.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K Ibrahim, Study Chair — Assiut University
Locations (1):
- Primary health care center, Asyut, Egypt